CLINICAL TRIAL: NCT03233776
Title: Safety and Efficacy of Interleukin-1 Inhibitor Anakinra for the Amelioration of Fever During Neutropenia and Mucositis in Patients With Multiple Myeloma Receiving an Autologous Stem Cell Transplantation After High-dose Melphalan
Brief Title: Anakinra: Safety and Efficacy in the Management of Fever During Neutropenia and Mucositis in ASCT
Acronym: AFFECT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: SC35
Record Dates: First submitted 2017-07-19; First posted 2017-07-31 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2020-11

CONDITIONS: Multiple Myeloma
Keywords: Anakinra; Mucositis; Hematopoietic stem cell transplantation; Febrile neutropenia
MeSH Terms: conditions — Multiple Myeloma; Mucositis; Febrile Neutropenia | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: 3+3 design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anakinra (Experimental): Dosage form: intravenous. Dosage: either 100 mg, 200 mg or 300 mg. Frequency: once daily. Duration: 15 days (day -2 until day +12).
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Subjects will be treated with a daily dose of anakinra, intravenously, starting on day -2, until day +12 (day 0 is day of SCT). Predefined doses are 100 mg , 200 mg and 300 mg.
  Other Names: Kineret

SUMMARY:
Oral and intestinal mucositis are major risk factors for the occurrence of fever during neutropenia and bloodstream infections after intensive chemo- and radiotherapy. These complications often require dose reductions or cause delay of treatment, and thereby interfere with optimal anticancer treatment. Currently, there are no effective strategies to prevent or treat mucositis and the related complications.

The pro-inflammatory cytokine interleukin-1β (IL-1β) has shown pivotal in the pathogenesis of mucositis and recently, it has been established in murine models that IL-1 inhibition significantly ameliorates chemotherapy-induced intestinal mucositis.

In this phase IIa study the safety, maximum tolerated dose and efficacy of anakinra, a recombinant human IL-1 receptor antagonist, will be determined in adult patients with multiple myeloma who receive high-dose melphalan (HDM) in the preparation for an autologous hematopoietic stem cell transplantation (ASCT) and are at high risk for experiencing mucositis and fever during neutropenia (FN). After establishing the optimal dose, a pivotal double-blind randomized placebo-controlled multicenter phase IIb trial will be planned to establish efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Diagnosed with multiple myeloma
* Scheduled to receive an autologous SCT after myeloablative therapy with high-dose melphalan
* Managed with a central venous catheter (triple- or quadruple lumen)
* Is able and willing to participate
* Has provided written informed consent
* Has a negative tuberculosis Quantiferon test
* Has negative serology for active hepatitis B and C
* Has negative serology for HIV
* Has no known hypersensitivity to Escherichia coli derived products or any components of anakinra
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation (during treatment with study medication), and for 30 days after the last dose.

Exclusion Criteria:

* Inability to understand the nature and extent of the trial and the procedures required
* Enrolment in any other investigational treatment study or use of an investigational agent during the stem cell transplantation (this means studies in multiple myeloma regarding induction or maintenance treatment are permitted).
* Women who are pregnant or nursing
* Diagnosed with amyloidosis or light-chain deposition disease
* ALT or AST greater than 2.0 x upper limit of normal (ULN) of the local laboratories values.
* Bilirubin levels greater than 2.0 x upper limit of normal (ULN) of the local Laboratories values, except for benign non-malignant indirect hyperbilirubinemia such as Gilbert syndrome
* Impaired renal function with eGFR <40 ml/min
* Received a live vaccine during the 3 months prior to baseline visit
* Recent use of IL-1 antagonist, such as anakinra, rilonacept or canakinumab, within three months prior to baseline visit
* Treatment with TNFα inhibiting agents (such as etanercept, adalimumab, infliximab, certolizumab and golimumab).
* Uncontrolled bacterial or viral infections, or fungal infections, at the start of therapy
* Documented colonization with highly resistant microorganisms (HRMOs, in Dutch: BRMO's), prior to registration, or detected during screening procedures
* Documented colonization with methicillin-resistant Staphylococcus aureus (MRSA), prior to registration
* Subjects who are not able to receive antibacterial prophylaxis with quinolones (because of hypersensitivity)
* Subjects with an active solid malignancy prior to registration, with the exception of cutaneous basal or squamous cell carcinomas
* History of mycobacterial infection.
* Subjects with intrinsic disorders of the gastro-intestinal (GI) tract, including, but not limited to: Crohn's disease, ulcerative colitis, celiac disease, short bowel syndrome.
* Subject has any concurrent medical or psychiatric condition or disease that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose of anakinra (MTD, 100, 200 or 300 mg). | Day of admission (day -2) until discharge. Maximum period: +30 days.
  In this study, using a traditional 3+3 design, 3 doses of anakinra will be examined: 100, 200 and 300 mg. The first cohort of patients will start with 100 mg. Escalation to the next dose cohort(s) is based on the occurrence of dose limiting toxicities (DLTs). The definition of a DLT is: an opportunistic infection, a SUSAR, severe non-hematological toxicity grade 3-4, or the occurrence of primary graft failure or prolonged neutropenia (neutrophils have not been >0.5 x10^9/l on one single day, assessed on day +21, and counting from day 0).

SECONDARY OUTCOMES:
Incidence of fever during neutropenia | Day of admission (day -2) until discharge. Maximum period: +30 days.
Incidence of mucositis-related fever | Day of admission (day -2) until discharge. Maximum period: +30 days.
Daily mean CRP level | Day of admission (day -2) until discharge. Maximum period: +30 days.
Intestinal mucositis as measured by the area-under-the-curve of reciprocal citrulline levels | Day of admission (day -2) until discharge. Maximum period: +30 days.
Clinical mucositis as determined by the daily mouth and gut scores | Day of admission (day -2) until discharge. Maximum period: +30 days.
Days with fever (≥ 38.5° C) | Day of admission (day -2) until discharge. Maximum period: +30 days.
Incidence of bloodstream infections i.e. bacteremia | Day of admission (day -2) until discharge. Maximum period: +30 days.
Length of hospital stay in days | Day of admission (day -2) until discharge. Maximum period: +30 days.
Use of systemic antimicrobial agents (incidence and duration) | Day of admission (day -2) until discharge. Maximum period: +30 days.
Use of analgesic drugs (incidence and duration) | Day of admission (day -2) until discharge. Maximum period: +30 days.
Use of total parenteral nutrition (TPN) (incidence and duration) | Day of admission (day -2) until discharge. Maximum period: +30 days.
Quality of life | Baseline, at discharge (average: 23 days; maximum: after 30 days), +100 days, +1 year
  Quality of life according to the EORTC QLQ-C30
Fatigue severity | Baseline, at discharge (average: 23 days; maximum: after 30 days), +100 days, +1 year
  Severity of fatigue as the score measured by the validated FACIT-Fatigue scale
Short term overall survival | +100 days and +1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Blijlevens, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

REFERENCES:
- [Derived] Wardill HR, de Mooij CEM, Da Silva Ferreira AR, Havinga H, Harmsen HJM, van der Velden WJFM, van Groningen LFJ, Tissing WJE, Blijlevens NMA. Supporting the gastrointestinal microenvironment during high-dose chemotherapy and stem cell transplantation by inhibiting IL-1 signaling with anakinra. Sci Rep. 2022 May 11;12(1):6803. doi: 10.1038/s41598-022-10700-3. PMID 35546555